CLINICAL TRIAL: NCT01902888
Title: Retrospective Evaluation of the GORE® VIABAHN® Endoprosthesis for a Popliteal Artery Aneurysm Indication
Brief Title: Evaluation of GORE® VIABAHN® Endoprosthesis for Popliteal Artery Aneurysm
Acronym: PAA 12-01
Status: Terminated | Type: Observational
Why Stopped: Closed due to internal and external factors.
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: PAA 12-01
Record Dates: First submitted 2013-07-16; First posted 2013-07-18 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Popliteal Artery Aneurysm
Keywords: popliteal artery; aneurysm; popliteal artery aneurysm; asymptomatic aneurysm; mural thrombus; Viabahn; Gore; Endoprosthesis
MeSH Terms: conditions — Popliteal Artery Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Popliteal aneurysm: GORE® VIABAHN® Endoprosthesis used to treat popliteal aneurysm
  Interventions: Device: GORE® VIABAHN® Endoprosthesis

INTERVENTIONS:
Device: GORE® VIABAHN® Endoprosthesis
  Other Names: Viabahn

SUMMARY:
This is a multicenter, non-randomized, single arm, retrospective study of GORE® VIABAHN® Endoprosthesis for the treatment of a Popliteal Artery Aneurysm (PAA).

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety and efficacy of the GORE® VIABAHN® Endoprosthesis for the treatment of subjects with Popliteal Artery Aneurysms. The study population includes subjects with an asymptomatic aneurysm (≥ 2 cm diameter) of the popliteal artery, symptomatic aneurysm (no diameter requirement) of the popliteal artery, or presence of mural thrombus (no diameter requirement) of the popliteal artery treated with the GORE® VIABAHN® Endoprosthesis between January 1, 2002 and December 31, 2010. Starting with most recently treated within the above date range, patients meeting Inclusion/Exclusion will be enrolled, until a minimum of 50 subjects with adequate follow up to determine primary endpoints through 12 months will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Received a GORE® VIABAHN® Endoprosthesis between January 1, 2002 and December 31, 2010 to treat a popliteal artery aneurysm;
* Had an asymptomatic aneurysm (≥ 2 cm diameter) of the popliteal artery, or symptomatic aneurysm (no diameter requirement) of the popliteal artery, or the presence of mural thrombus (no diameter requirement) of the popliteal artery;
* Was 18 years of age or older; and
* Had an elective popliteal artery aneurysm procedure.

Exclusion Criteria:

* Bilateral popliteal artery aneurysms with initial treatment on the same day
* Had previous surgery for the popliteal artery aneurysm in the study limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had popliteam aneurysm and were treated with GORE® VIABAHN® Endoprosthesis between January 1, 2002 and December 31, 2010.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hector Novoa, BS, Study Director — W. L. Gore & Associates, Inc (sponsor)
Locations (3):
- United States (3):
  - Baptist Health, Miami, Florida
  - The Vascular Group of Naples, Naples, Florida
  - Washington University School of Medicine, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Groups:
- Popliteal Aneurysm: GORE® VIABAHN® Endoprosthesis used to treat popliteal aneurysm
  GORE® VIABAHN® Endoprosthesis
Period: Overall Study
Arm/Group | Popliteal Aneurysm
Started | 3
Completed | 0
Not Completed | 3
Not completed — Study Terminated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Popliteal Aneurysm
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: The Number of Patients That do Not Have a Failure of Technical Success or Loss of Primary Patency.
Description: A composite of freedom from failure of technical success or loss of primary patency at 12 months
Time Frame: 12 months following initial study procedure
Arm/Group | Popliteal Aneurysm
Number analyzed (Participants) | 0

2. Primary Outcome: Primary Safety Endpoint: Number of Serious Adverse Events (Related to Initial Procedure or the Device Itself) That Occur Within 30 Days of the Initial Study Procedure.
Description: 30 day serious adverse events related to the initial study procedure or the study device.
Time Frame: 30 days following initial study procedure
Arm/Group | Popliteal Aneurysm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Popliteal Aneurysm
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination of study. No subject analysis done

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No